CLINICAL TRIAL: NCT01159327
Title: A Randomized Phase II Study of Sorafenib Maintenance in Patients With Extensive Disease Small Cell Lung Cancer (ED-SCLC) After Response to Induction Chemotherapy
Brief Title: Study of Sorafenib Maintenance in Patients With ED-SCLC After Response to Induction Chemotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrolling participants
Sponsor: National Cancer Center, Korea (Other Government)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ji-youn Han, Head, Center for Lung Cancer, National Cancer Center, Korea
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCCTS-10-476
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2015-11-11 (Estimated); Status verified 2015-11

CONDITIONS: Small Cell Lung Cancer
Keywords: Sorafenib (nexavar); ED-SCLC; Maintenance; Extensive Disease Small cell lung cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm A (Experimental): Sorafenib maintenance arm
  Interventions: Drug: Sorafenib
- Arm B (No Intervention): observation arm

INTERVENTIONS:
Drug: Sorafenib — Sorafenib 400mg, bid(800mg/day), daily, PO
  Other Names: Nexavar
  Arms: Arm A

SUMMARY:
A Phase I trial of weekly topotecan in combination with sorafenib in treatment of relapsed Small cell lung cancer (SCLC) has been commenced. In the present randomized phase 2 study, the investigators will research whether Sorafenib maintenance prolongs progression free survival (PFS) and overall survival (OS) in patients with ED-SCLC who achieved CR or PR after platinum-based induction chemotherapy.

DETAILED DESCRIPTION:
Small cell lung cancer (SCLC) comprises 10-15 % of all lung cancer. Despite high responsiveness to initial chemotherapy, its high relapse rate makes the treatment of SCLC is challenging. With platinum plus etoposide or irinotecan, overall response rate is as high as 85%, however, the median duration of response is short (approximately 4 months), and median survival times are 9 to 11 months, with a 2-year survival rate of less than 10% [J Clin oncology. 2009 Oct 1;27(28):4787-92]. New and more effective agents are clearly needed against SCLC. Sorafenib is a multikinase inhibitors acting on pathways involved in tumour progression and angiogenesis, and is undergoing investigation for the treatment of SCLC in either the first- or second-line setting. The only data available so far are on sorafenib, which seems to be a promising agent with a median survival of 7 and 5 months in platinum-sensitive and platinum-refractory patients, respectively (2008 J Clin oncology 26. Abstract 8039). This compared favourably with historical controls receiving salvage chemotherapy.

ELIGIBILITY:
Inclusion criteria:

* Histologically or cytologically confirmed ED-SCLC patients who have achieved a complete or partial response after four to six cycles of platinum based induction chemotherapy.
* Extensive stage SCLC is defined as disease not meaning the definition of limited stage disease
* Previous radiotherapy is allowed only if < 30% of marrow bearing bones were irradiated and if radiotherapy was completed at least 2 weeks prior to enrollment and the patient has recovered from all adverse effects of prior radiotherapy.
* Age >18 years.
* Written informed consent that is consistent with ICH-GCP guidelines
* Life expectancy of greater than 3 months.
* ECOG performance status 2 (Karnofsky ≥50%).
* Ability to swallow oral medication
* Women of childbearing potential must have a negative serum pregnancy test performed within 7 days prior to the start of treatment
* Both men and women enrolled in this trial must use adequate barrier birth control measures during the course of the trial and during the first 3 months after the completion of trial
* Adequate bone marrow, liver and renal function

Exclusion Criteria:

* History of cardiac disease/ HIV infection / chronic hepatitis B or C / of organ allograft
* Active clinically serious infections
* Patients with seizure disorder requiring medication or evidence or history of bleeding diathesis or coagulopathy
* Patients undergoing renal dialysis
* Pulmonary hemorrhage/ bleeding event ≥ CTCAE grade 2 within four weeks
* Any other hemorrhage/ bleeding event ≥ CTCAE grade 3 within four weeks
* Non-healing wound, ulcer or bone fracture
* Thrombotic or embolic venous or arterial events of study drug
* Previous or concurrent cancer that is distinct in histology of primary site, EXCEPT cervical carcinoma in situ, treated basal cell carcinoma, superficial bladder tumors (Ta, Tis, T1). Any cancer curatively treated >3 years prior to entry is permitted.
* Substance abuse, medical, psychological or social conditions that may interfere with the subject's participation in the study or evaluation of the study results
* Known or suspected allergy or any other contraindication for Sorafenib administration
* Pregnant or breast-feeding women.
* Any disease which could affect the evaluation of the study drug
* Any condition that is unstable or could jeopardize the safety of the subject and their compliance in the study
* Any condition which could affect the absorption or pharmacokinetics of the Study drug including any type of gastrointestinal resection or surgery
* Uncontrolled symptomatic brain metastasis

Excluded therapies and medications, previous and concomitant:

* Investigational drug or device therapy including outside of this trial during or within 4 weeks prior to study entry (signing Informed Consent).
* The toxicity effects of previous antitumor chemotherapy or immunotherapy must be resolved to less than CTC Grade 2 level (exception: alopecia).
* Prior treatment with other VEGFR inhibitors (i.e. sunitinib, thalidomide, vandetanib and other experimental agents of this class).
* Major surgery within 4 weeks prior to start of study (Informed Consent signature). Minimal invasive biopsy is allowed.
* Use of biologic response modifiers, such as G-CSF, within 3 weeks prior to study entry. [Therapeutic G-CSF and other hematopoietic growth factors may be used in the management of acute toxicity such as febrile neutropenia when clinically indicated or at the discretion of the investigator, however they may not be substituted for a required dose reduction].
* Any agents which could affect the absorption or pharmacokinetics of the study drug
* Prior exposure to the study drug
* Therapeutic anticoagulation with vitamin K antagonists such as warfarin, or with heparins or heparinoids. Prophylactic low dose warfarin (1 mg po qd) is permitted if the INR (International normalized ratio) is ≤ 1.5. Low-dose aspirin is permitted (80-100 mg daily).

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-12; Primary Completion 2013-04 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Progression-free survival | every 8 weeks
  Progression-free survival was calculated from the randomization date until evidence of PD or death

SECONDARY OUTCOMES:
Overall survival | the date of registration to the date of death
  The duration of overall survival is measured from randomization date to the date of death from any cause or the last follow-up examination
Toxicity | First drug intake until 30 days after last treatment admisitration
  For grading of adverse events CTCAE criteria (version 4.0) will be utilized. All adverse events occurring between first drug intake until 30 days after last treatment administration will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: JI-YOUN HAN, PhD.MD, Principal Investigator — National Cancer Center
Locations (1):
- National Cancer Center, Korea, Goyang-si, Gyeonggi-do, South Korea